CLINICAL TRIAL: NCT05334732
Title: Improving Communication and Adherence in Black Breast Cancer Survivors
Brief Title: Improving Communication and Adherence in Black Breast Cancer Survivors (Sisters Informing Sisters)
Acronym: SIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-19-15740; HM20016396 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Black Women; Breast Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sisters Informing Sisters Sessions (Experimental): The intervention is peer-based and in concert with our theoretical model, builds upon positive role-modeling of the survivor coach to the patient, addresses behavioral expectations/capacities, and uses Motivational Interviewing (MI) techniques. The intervention includes a culturally relevant coach's manual and a patient workbook that will be used to facilitate the coaching sessions.
  Interventions: Behavioral: SIS TALK Back Intervention
- Enhanced Usual Care (No Intervention): Women in the EUC arm will receive usual care that includes standardized information in the public domain (NCI treatment information booklet). This booklet was chosen to provide women with national-level recommendations regarding treatment recommendations.

INTERVENTIONS:
Behavioral: SIS TALK Back Intervention — The participants in this arm will be seen by a trained survivor coach and receive culturally tailored intervention materials.
  Arms: Sisters Informing Sisters Sessions

SUMMARY:
The purpose of this study is to test an evidence-based intervention designed to increase adherence to systemic therapy in Black women compared to enhanced usual care.

DETAILED DESCRIPTION:
Black women continue to experience worse breast cancer outcomes, which may be due to inadequate adherence to systemic therapies that can be improved via patient-centered communication. We developed and piloted the Sisters Informing SistersSM (SIS) intervention (survivor-led skill-building sessions and culturally tailored materials to activate Black breast cancer survivors in their medical encounters) and obtained promising findings. This project will compare in a two-arm RCT the impact of SIS vs. enhanced usual care (treatment recommendation summary form) on patient-centered communication and systemic treatment adherence; SIS tools may be integrated within existing clinical and support services.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black
* Newly diagnosed (~4 weeks post-definitive surgery and prior to initiation of adjuvant chemotherapy or endocrine therapy) patients (stage I-III)
* Eligible for chemotherapy or endocrine therapy according to NCCN guidelines, but have not initiated systemic therapy
* Ability to read and speak English
* Ability to provide meaningful consent as determined by trained study personnel and/or a member of the patient's care team
* No prior cancer treatment (other than skin cancer) in the two years preceding enrollment
* Physicians Must be a license doctor of study patient(s)
* Ability to speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Assessing Study Adherence Behaviors- Initiation | 36 Months
  Initiation will be measured for all therapies based on the number of participants starting at least one cycle of prescribed therapy
Assessing Study Adherence Behaviors- Delay of Adjuvant or Endocrine Therapy. | 36 Months
  Initiation Delay of therapy will be measured by the number of participant's days from definitive surgery date to the date of her first cycle of adjuvant systemic therapy. Classifications of delay are dichotomized according to published reports (<60 days primary measure).
Assessing Study Adherence Behaviors- Overall Chemotherapy Adherence | 36 Months
  Overall chemotherapy adherence will be measured by the number of participants that complete chemotherapy. Chemotherapy adherence will be measured as having at least 80% or more of the recommended doses. Adherence will be calculated based on the planned and expected number of cycles divided by the number received (i.e., 6 chemotherapy cycles received/8 expected = 75% adherent).

SECONDARY OUTCOMES:
Assess Perceived Involvement in Care: PCC Outcomes - Level of Engagement in Decision Making | 36 Months
  The number of participants level of engagement in decision-making will be assessed by utilizing The Perceived Involvement in Care (PCC) 13-Item scale. PCC will be assessed via direct observation of medical encounters through a quantitative analysis of audiotaped visits.
Assess Perceived Involvement in Care: PCC Outcomes - Perceptions of Doctor Behaviors by determining a more patient-centered encounter vs a more biomedically focused encounter. | 36 Months
  The number of participants level of engagement in perceptions of doctor behaviors will be assessed by utilizing The Perceived Involvement in Care (PCC) 13-Item scale. PCC will be assessed via direct observation of medical encounters through a quantitative analysis of audiotaped visits. A value >1 indicates a more patient-centered encounter, whereas a value <1 indicates a more biomedically focused encounter.
Assess Perceived Involvement in Care: PCC Outcomes - Perceptions of Patient Behaviors by determining Perceptions of Doctor Behaviors by determining a more patient-centered encounter vs a more biomedically focused encounter | 36 Months
  The number of participants level of engagement in perceptions of patient behaviors will be assessed by utilizing The Perceived Involvement in Care (PCC) 13-Item scale. PCC will be assessed via direct observation of medical encounters through a quantitative analysis of audiotaped visits. A value >1 indicates a more patient-centered encounter, whereas a value <1 indicates a more biomedically focused encounter.
Determine Process and Implementation Outcomes | 36 Months
  Assess the number of participants who Consent to Participate in the trial
Determine Process and Implementation Outcomes | 36 Months
  Assess the number of participants that participate in the trial after they sign consent
Determine Process and Implementation Outcomes | 36 Months
  Assess the Cost of the trial per arm. Personnel time costs will be obtained by multiplying the staff time. costs by hourly average wage and fringe benefit rates. The staff time will include the training to identify at-risk women and the time spent administering/reviewing study materials including the treatment summary request form

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa B Sheppard, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.